CLINICAL TRIAL: NCT06175338
Title: Randomized Double Blind Phase I Trial Comparing Pharmacokinetics, Pharmacodynamics, Immunogenicity and Safety of Rituximab (Mabscale LLC, Russia)+ Methotrexate+ Folic Acid and MabThera® Methotrexate+ Folic Acid in Adult Patients With Moderate or Severe Rheumatoid Arthritis With Insufficient Response to Treatment Tumor Necrosis Factor (TNF-α)
Brief Title: Study, Evaluating Pharmacokinetics, Pharmacodynamics, Immunogenicity and Safety Profiles of Rituximab Compared to MabThera® in Patients With Rheumatoid Arthritis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mabscale, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RIT-1/01092021
Record Dates: First submitted 2023-12-07; First posted 2023-12-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab (manufactured by Mabscale, LLC) (Experimental): Eligible subjects (104 patients) will receive Rituximab 1000 mg in 150 ml 0,9 % NaCl (total volume of infusion 250 ml) twice: on Visit 1 and 5. The following visits are the visits of safety and PK, PD and immunogenicity and also preliminary effectiveness). Patients will also receive background treatment Methotrexate+ Folic acid.
  Interventions: Drug: Rituximab
- MabThera® (Active Comparator): Eligible subjects (104 patients) will receive MabThera® 1000 mg in 150 ml 0,9 % NaCl (total volume of infusion 250 ml) twice: on Visit 1 and 5. The following visits are the visits of safety and PK, PD and immunogenicity and also preliminary effectiveness). Patients will also receive background treatment Methotrexate+ Folic acid.
  Interventions: Drug: MabThera®

INTERVENTIONS:
Drug: Rituximab — Rituximab 1000 mg in 150 ml 0,9 % NaCl (total volume of infusion 250 ml)
  Arms: Rituximab (manufactured by Mabscale, LLC)
Drug: MabThera® — MabThera® 1000 mg in 150 ml 0,9 % NaCl (total volume of infusion 250 ml)
  Arms: MabThera®

SUMMARY:
A randomised, double blind, parallel group, multicentre study to compare the pharmacokinetics, pharmacodynamics, immunogenicity and safety of Rituximab (Mabscale LLC, Russia) versus MabThera® in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
RIT-1/01092021 is a double-blind randomized, parallel group, multicenter clinical trial comparing pharmacokinetics, pharmacodynamics, immunogenicity and safety of Rituximab (Mabscale LLC, Russia) and MabThera® in adult patients with moderate or severe rheumatoid arthritis with insufficient response to treatment tumor necrosis factor (TNF-α) inhibitors receiving background treatment with methotrexate. The purpose of the study is to demonstrate equivalence of pharmacokinetics, pharmacodynamics, immunogenicity and safety of Rituximab (Mabscale LLC, Russia) and MabThera®. The study will take place across approximately 30 study sites in Russia in order to randomize 208 patients. Rituximab is a monoclonal antibody currently being developed by Mabscale LLC, as a proposed biosimilar to MabThera®, which is approved as treatment in case of insufficient response or toxicity to treatment tumor necrosis factor (TNF-α) inhibitors receiving background treatment with methotrexate. This randomized equivalence study is designed to meet the regulatory requirement for approval of a biosimilar product.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female 18-65 y.o. with body weight 50-120 kg
* Patients with active rheumatoid arthritis with disease duration minimum 6 months prior to screening visit per ACR/EULAR 2019 criteria classification.
* Moderate or severe active course of rheumatoid arthritis, which is defined as the fulfillment of all of the following conditions:

  * ≥6 tender joints (based on a score of 68 joints) at screening and baseline; And
  * ≥6 swollen joints (based on a score of 66 joints) at screening and at baseline; And
  * level of C-reactive protein is not less than 10 mg/l or ESR is not less than 28 mm/hour at screening.
* Positive result of the analysis for antibodies to cyclic citrullinated peptide (≥10 units/ml) and / or the presence of rheumatoid factor (≥ 20 units/ml) at screening (see section).
* Received treatment for RA and experienced an inadequate response or intolerance to treatment with at least 1 anti-TNF alpha therapy;
* Must have received MTX for a minimum of 12 weeks, with the last 4 weeks, prior to screening at a stable dose 10-25 mg/week;

Exclusion Criteria:

* Contraindications according to the MabThera SmPC and every serious coexisting diseases which, in the Investigator's opinion, would preclude subject participation
* History of current rheumatic autoimmune disease other than RA and current inflammatory joint disease other than RA
* Positive tests for HIV, hepatitis B surface antigen (HBsAg) Anti-HBc antibody, hepatitis C antibody
* Prior treatment with rituximab, other anti-CD20 mAb
* Pregnancy or lactation or women planning to get pregnant during the course of the study and/or within 12 months post last study drug infusion
* COVID prior 8 weeks prior to Screening visit or other acute systemic infection within 4 weeks prior to Day 1
* Allergic reaction or intolerance to rituximab, MabionCD20 or any of their components
* Severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or previous treatment of any lymphocyte-depleting therapies
* Confirmed current active tuberculosis (TB).
* Any significant cardiac disease
* History of a severe allergic reaction or anaphylactic reaction to a biological agent or history of hypersensitivity to any component of the study drug including known hypersensitivity or allergy to a murine product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
AUC(w2-24) | Day 1 to Week 24
  Area Under the Concentration Time Curve predose Day 1 to Week 24 (AUC(w2-24).
AUC0-inf | Day 1 to Week 24
  Area Under the Concentration Time Curve extrapolated from 0 to infinity (AUC0-inf)
Cmax | Dose 2 to the end of the study or Week 24
  Maximum Plasma Concentration (Cmax) after Dose 2

SECONDARY OUTCOMES:
Ctrough | Day 1 to Day 15
  Residual concentration (Ctrough) before the second infusion on Day 15
AUC0-d15 | Day 1 - Day 15 (before infusion)
  Area under the concentration-time curve from 0 (directly pre-infusion on Day 1) before pre-infusion measurement on Day 15 (AUC0-d15)
AUC0-w12 | Day 1 - Week 12 (before infusion)
  Area under the concentration-time curve from 0 and before measurement at Week 12 (AUC0-w12)
AUCd15-n24 | Day 15 - Week 24
  Area under the concentration-time curve from measurement immediately before the second infusion (Day 15) before measuring in point Week 24 (AUCd15-n24)

CONTACTS AND LOCATIONS:
Locations (12):
- Russia (12):
  - Immanuel Kant Baltic Federal University, Kaliningrad
  - Scientific-Research Medical Complex Your Health, Kazan'
  - LLC "Medical Center Revma-Med", Kemerovo
  - LLC "Korolev Family Clinic №4", Korolyov
  - Moscow City Clinical Hospital №1, Moscow
  - V.A. Nasonova Research Institute of Rheumatology, Moscow
  - Orenburg State Medical University, Orenburg
  - JSC "Northwestern Center for Evidence-Based Medicine", Saint Petersburg
  - LLC "Interleukin", Saint Petersburg
  - Medical center "Capital-Polis", Saint Petersburg
  - Saratov State Medical University, Saratov
  - LLC "Biomed", Vladimir

IPD SHARING:
Plan to Share IPD: No